CLINICAL TRIAL: NCT04071587
Title: Brain Computer Interface Training for Patients With Severe Upper Limb Paresis in the Subacute Phase After Stroke
Brief Title: Brain Computer Interface Training After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Hammel Neurorehabilitation Centre and University Research Clinic (Other); Sygekassernes Helsefond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 649780
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-01

CONDITIONS: Stroke
Keywords: BCI; upper limb; severe paresis; subacute stroke; rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: Patients are randomized to one of two treatment options, intervention or standard rehabilitation
Who Masked: Outcomes Assessor
Masking Description: All assessments will be done by assessors blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCI training (Experimental): Patients randomized to this group will receive up to12 (minimum 8) sessions of BCI training with the RecoveriX system (gtec, Austria). The system combines EEG driven functional electrical stimulation with visual feedback. BCI training is provided as a part of standard training of the impaired upper limb.
  Interventions: Device: Brain Computer Interface training
- Control (Active Comparator): Patients randomized to this control group will receive standard physiotherapy and occupational therapy for their impaired upper limb.
  Interventions: Behavioral: Control

INTERVENTIONS:
Device: Brain Computer Interface training — Training with RecoveriX system.
  Arms: BCI training
Behavioral: Control — Standard physiotherapy and occupational therapy according to clinical routines.
  Arms: Control

SUMMARY:
In this study, we want to examine the effect of a new treatment approach for patients with severe upper limb paresis in the subacute phase after stroke. Brain Computer Interface (BCI) driven functional electrical stimulation will be compared to conventional training.

DETAILED DESCRIPTION:
A randomized controlled pilot study will be conducted. Forty patients with severe UL paresis will be included. Patients with severe hemiparesis after stroke will be allocated to one of two treatment groups by a computerized randomization program. Patients in the intervention group will receive training with a BCI system paired with functional electrical stimulation and visual feedback (RecoveriX, gtec, Austria) as part of their rehabilitation. The targeted number of training sessions in the intervention group is 12. Patients in the control group will receive conventional upper limb training. All patients will receive other rehabilitation according to their needs.

Patients will be assessed by blinded raters before and after the intervention and 3 months post stroke. Main endpoint will be UL motor function assessed by Action Research Arm Test (ARAT) at 3 months post stroke. Other outcome measures comprise Fugl Meyer Motor Assessment and Functional Independence Measure. The patients and therapists' experience with this type of training will be evaluated with questionnaires and interviews.

ELIGIBILITY:
Inclusion Criteria:

* First ever or former stroke without UL motor residuals as confirmed by CT and / or MRI
* 15 days to 60 days (+/- 3) after stroke onset
* Severe paresis or paralysis defined as < 13 on Action Research arm Test (ARAT)
* Able to give informed consent
* Able to comply with treatment protocol.

Exclusion Criteria:

* Other conditions limiting functional use of the affected UL,
* Psychiatric / behavioral conditions that interfere with compliance to the protocol, epilepsy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Upper limb function 90 days after stroke
  Upper limb function on a scale of 0 - 57 (best)

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (UL) | Upper limb impairment 90 days after stroke
  Upper limb impairment on a scale from 0-66 (best)
Functional Independence Measure | Functional independence 90 days after stroke
  Independence in activities og daily living, 18-126 (best)

OTHER OUTCOMES:
Interviews | Through study completion, an average of 6 months
  Qualitative assessment of user experiences

CONTACTS AND LOCATIONS:
Overall Officials: Iris Brunner, PhD, Principal Investigator — Aarhus University, Hammel Neurocenter
Locations (1):
- Hammel Neurorehabilitation Centre and University Research Clinic, Hammel, Aarhus, Denmark